CLINICAL TRIAL: NCT00691301
Title: A Limited Access Phase II Trial of Pemetrexed (Alimta, LY231514) (NSC #698037) in Combination With Cisplatin (NSC #119875) in the Treatment of Advanced, Persistent, or Recurrent Carcinoma of the Cervix
Brief Title: Pemetrexed and Cisplatin in Treating Patients With Advanced, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0076GG; GOG-0076GG; CDR0000597154 (Other: CDR); NCI-2009-00572 (Other: NCI)
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2015-05

CONDITIONS: Cervical Cancer
Keywords: cervical squamous cell carcinoma; recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed and cisplatin (Experimental): Pemtrexed plus cisplatin on day 1 every 21 days
  Interventions: Drug: cisplatin; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: cisplatin — Cisplatin as an IV infusion at less than 1 mg/min over less than 4 hours at a dose of
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed together with cisplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving pemetrexed together with cisplatin and to see how well it works in treating patients with advanced, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the antitumor activity of pemetrexed disodium and cisplatin with objective tumor response (partial and complete response) in patients with advanced, persistent, or recurrent carcinoma of the cervix.
* To determine the nature and degree of toxicity of this regimen in these patients.

Secondary

* To determine the effects of this regimen on progression-free survival and overall survival.

OUTLINE: This is a multicenter study. Patients are stratified according to prior cisplatin therapy as a radiosensitizer (yes vs no).

Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 1-4 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous or nonsquamous cell carcinoma of the cervix

  * Advanced, persistent, or recurrent disease
* Disease not amenable to curative therapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have ≥ 1 target lesion to be used to assess response

  * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days following completion of radiotherapy

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Platelet count ≥ 100,000/mm^3
* ANC ≥ 1,500/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 60 mL/min
* SGOT ≤ 2.5 times ULN (≤ 5 times ULN if due to hepatic metastases)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN if due to hepatic metastases)
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neuropathy (sensory and motor) ≤ grade 1
* Able to take folic acid, vitamin B12, and dexamethasone according to study protocol
* No history of other invasive malignancies within the past 5 years, except nonmelanoma skin cancer
* No active infection requiring antibiotics with the exception of uncomplicated UTI
* No presence of third space fluid which cannot be controlled by drainage

PRIOR CONCURRENT THERAPY:

* Recovered from effects of recent surgery, radiotherapy, or other therapy
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* At least 4 weeks since prior radiotherapy
* More than 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin and patient remains free of recurrent or metastatic disease
* No prior radiotherapy to any portion of the abdominal cavity or pelvis except for the treatment of cervical cancer
* No prior radiotherapy to more than 25% of marrow-bearing areas
* No prior cancer treatment that contraindicates study treatment
* No prior cytotoxic drugs for advanced or recurrent carcinoma of the cervix

  * Prior cisplatin as a radiosensitizer for primary treatment of disease allowed
* No nonsteroidal anti-inflammatory drugs (NSAIDs) or salicylates 2-5 days before, during, or for 2 days after receiving pemetrexed disodium

  * No NSAIDS with a long half-life (e.g., naproxen, piroxicam, diflunisal, or nabumetone) 5 days before, during, and for 2 days after receiving pemetrexed disodium
* Concurrent hormone replacement therapy is permitted
* Concurrent daily low-dose acetylsalicylic acid therapy (≤ 325 mg/day) allowed
* Concurrent use of acetylsalicylic acid (up to 1.3 g/day) allowed

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (12):
- United States (12):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Women's Cancer Center - La Canada, Las Vegas, Nevada
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Saint Francis Campus, Tulsa, Oklahoma
  - Parkland Memorial Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed and Cisplatin: Pemtrexed plus cisplatin on day 1 every 21 days
  cisplatin: Cisplatin as an IV infusion at less than 1 mg/min over less than 4 hours at a dose of
  pemetrexed disodium
Period: Overall Study
Arm/Group | Pemetrexed and Cisplatin
Started | 55
Completed | 1
Not Completed | 54
Not completed — Adverse Event | 10
Not completed — Death | 2
Not completed — Lack of Efficacy | 32
Not completed — Withdrawal by Subject | 4
Not completed — Concurrent illness | 2
Not completed — other reason | 3
Not completed — Did not initiate study treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed and Cisplatin
Number analyzed (Participants) | 54
Age, Customized [Number; unit: participants]
  20-29 years | 3
  30-39 years | 10
  40-49 years | 23
  50-59 years | 15
  >60 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 29
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle until disease progression or study withdrawal; and at any other time if clinically indicated, up to 5 years.
Population: Individuals who initiated study treatment
Measure: Number; unit: participants
Arm/Group | Pemetrexed and Cisplatin
Number analyzed (Participants) | 54
participants
  Complete Response | 1
  Partial Response | 16

2. Primary Outcome: Frequency and Severity of Observed Adverse Effects
Description: All eligible and evaluable patients
Time Frame: every 21 days during study treatment and up to 30 days after the last cycle of treatment.
Population: All eligible and evaluable patients.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
Participants
  Leukopenia | 16 | 8 | 15 | 12 | 3 | 0
  Thrombocytopenia | 32 | 11 | 5 | 3 | 3 | 0
  Neutropenia | 20 | 5 | 10 | 12 | 7 | 0
  Anemia | 2 | 17 | 22 | 6 | 7 | 0
  Other hematologic | 49 | 0 | 3 | 1 | 1 | 0
  Allergy/immunology | 49 | 3 | 0 | 1 | 1 | 0
  Auditory/ear | 39 | 0 | 14 | 1 | 0 | 0
  Cardiac | 47 | 5 | 2 | 0 | 0 | 0
  Coagulation | 53 | 0 | 0 | 1 | 0 | 0
  Constitutional | 6 | 12 | 23 | 12 | 1 | 0
  Dermatologic | 24 | 20 | 9 | 1 | 0 | 0
  Endocrine | 53 | 1 | 0 | 0 | 0 | 0
  Nausea | 7 | 19 | 22 | 6 | 0 | 0
  Vomiting | 19 | 11 | 17 | 7 | 0 | 0
  Gastrointestinal | 4 | 15 | 24 | 10 | 1 | 0
  Genitourinary/renal | 43 | 6 | 4 | 1 | 0 | 0
  Hemorrhage | 44 | 7 | 0 | 2 | 1 | 0
  Infection | 37 | 0 | 11 | 6 | 0 | 0
  Lymphatics | 42 | 5 | 7 | 0 | 0 | 0
  Metabolic | 10 | 19 | 10 | 10 | 5 | 0
  Musculoskeletal | 50 | 3 | 0 | 1 | 0 | 0
  Neurosensory | 31 | 15 | 6 | 2 | 0 | 0
  Other neurological | 42 | 8 | 3 | 1 | 0 | 0
  Ocular/visual | 44 | 6 | 2 | 2 | 0 | 0
  Pain | 18 | 11 | 13 | 12 | 0 | 0
  Pulmonary | 37 | 9 | 6 | 2 | 0 | 0
  Sexual/reproductive | 53 | 1 | 0 | 0 | 0 | 0
  Syndromes | 52 | 1 | 1 | 0 | 0 | 0
  Vascular | 50 | 0 | 3 | 1 | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Duration of progression-free survival in months.
Time Frame: From enrollment onto the study until the onset of disease progression or death, up to 5 years
Population: Individuals who initiated study treatment
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pemetrexed and Cisplatin
Number analyzed (Participants) | 54
months | 5.6 [2.6 to 9.0]

4. Secondary Outcome: Duration of Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually, up to 5 years.
Population: Eligible and treated patients
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed and Cisplatin
Number analyzed (Participants) | 54
months | 12.3 [0.3 to 38.6]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Pemetrexed and Cisplatin
Serious Adverse Events (participants affected / at risk) | 23/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Cisplatin (N=54)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Death No Ctcae Term - Sudden Death (General disorders) | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1
Perforation, Gi - Appendix (Gastrointestinal disorders) | 1
Perforation, Gi - Colon (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 3
Hemorrhage, Gi - Stomach (Vascular disorders) | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 1
Febrile Neutropenia (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 2
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Pain: Chest Wall (General disorders) | 1
Pain: Head/Headache (General disorders) | 1
Pain: Back (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 3
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Cisplatin (N=54)
Allergy/Immunology - Other (Immune system disorders) | 2
Allergic Reaction/Hypersensitivity (Immune system disorders) | 3
Rhinitis (Immune system disorders) | 2
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 14
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 34
Platelets (Blood and lymphatic system disorders) | 22
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 38
Lymphopenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 52
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 3
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 5
Pericardial Effusion (Cardiac disorders) | 1
Inr (Vascular disorders) | 1
Ptt (Vascular disorders) | 1
Constitutional Symptoms - Other (General disorders) | 3
Sweating (General disorders) | 16
Weight Gain (General disorders) | 2
Fever (General disorders) | 16
Weight Loss (General disorders) | 4
Obesity (General disorders) | 1
Rigors/Chills (General disorders) | 11
Fatigue (General disorders) | 47
Insomnia (General disorders) | 10
Nail Changes (Skin and subcutaneous tissue disorders) | 2
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 17
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Decubitus (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7
Flushing (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hot Flashes (Endocrine disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 4
Dental: Teeth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 7
Taste Alteration (Gastrointestinal disorders) | 9
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 7
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Necrosis, Gi - Stoma (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Anus (Gastrointestinal disorders) | 2
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 13
Mucositis (Clinical Exam) - Esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 35
Anorexia (Gastrointestinal disorders) | 33
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 47
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 26
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 9
Hemorrhage, Gi - Rectum (Vascular disorders) | 8
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hemorrhage, Gi - Anus (Vascular disorders) | 1
Hemorrhage, Gu - Uterus (Vascular disorders) | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1
Hemorrhage, Gu - Kidney (Vascular disorders) | 1
Hemorrhage, Gi - Stomach (Vascular disorders) | 1
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Salivary Gland (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 13
Infection - Other (Infections and infestations) | 1
Inf Unknown Anc: Vagina (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 3
Inf Unknown Anc: Salivary Gland (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2
Edema: Limb (Blood and lymphatic system disorders) | 15
Edema: Head And Neck (Blood and lymphatic system disorders) | 3
Ast (Metabolism and nutrition disorders) | 12
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 3
Proteinuria (Metabolism and nutrition disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 21
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Alt (Metabolism and nutrition disorders) | 11
Alkaline Phosphatase (Metabolism and nutrition disorders) | 15
Bilirubin (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 20
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 32
Hypokalemia (Metabolism and nutrition disorders) | 20
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 4
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 15
Mood Alteration - Anxiety (Nervous system disorders) | 11
Mood Alteration - Agitation (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Neuropathy-Sensory (Nervous system disorders) | 25
Neuropathy-Motor (Nervous system disorders) | 2
Ocular/Visual - Other (Eye disorders) | 1
Watery Eye (Eye disorders) | 2
Dry Eye (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Blurred Vision (Eye disorders) | 9
Pain - Other (General disorders) | 11
Pain: Urethra (General disorders) | 1
Pain: Pelvis (General disorders) | 8
Pain: Chest /Thorax Nos (General disorders) | 2
Pain: Chest Wall (General disorders) | 5
Pain: Throat/Pharynx/Larynx (General disorders) | 4
Pain: Head/Headache (General disorders) | 25
Pain: Neck (General disorders) | 4
Pain: Extremity-Limb (General disorders) | 13
Pain: Buttock (General disorders) | 2
Pain: Back (General disorders) | 18
Pain: Joint (General disorders) | 6
Pain: Bone (General disorders) | 3
Pain: Lymph Node (General disorders) | 2
Pain: Kidney (General disorders) | 1
Pain: Bladder (General disorders) | 1
Pain: Pain Nos (General disorders) | 1
Pain: Stomach (General disorders) | 2
Pain: Rectum (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 17
Pain: Oral - Gums (General disorders) | 1
Pain: Middle Ear (General disorders) | 1
Pain: External Ear (General disorders) | 3
Pain: Cardiac/ Heart (General disorders) | 2
Pain: Muscle (General disorders) | 3
Pain: Anus (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dlco (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21
Renal/Genitourinary - Other (Renal and urinary disorders) | 4
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 4
Incontinence, Urinary (Renal and urinary disorders) | 3
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 10
Vaginal Discharge (Reproductive system and breast disorders) | 5
Syndromes - Other (General disorders) | 1
Cytokine Release Syndrome (General disorders) | 2
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No